CLINICAL TRIAL: NCT01952574
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AMG 334 in Migraine Prevention
Brief Title: Study to Evaluate the Efficacy and Safety of Erenumab (AMG 334) in Migraine Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120178; 2012-005331-90 (EudraCT Number)
Record Dates: First submitted 2013-08-30; First posted 2013-09-30 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Migraine
Keywords: migraine, headache, prevention, prophylaxis
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Intervention Model Description: In the DBTP participants were randomized to one of four arms. In the optional CHU substudy participants were randomized into one of two treatment groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection during the double-blind treatment phase.
  In the open-label treatment phase participants received 70 mg erenumab QM from week 12 to week 264 (last dose). After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
  Interventions: Drug: Erenumab; Drug: Placebo
- Erenumab 7 mg QM (Experimental): Participants received erenumab 7 mg on day 1 and at weeks 4 and 8 by subcutaneous injection during the double-blind treatment phase.
  In the open-label treatment phase participants received 70 mg erenumab QM from week 12 to week 264 (last dose). After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
  Interventions: Drug: Erenumab
- Erenumab 21 mg QM (Experimental): Participants received erenumab 21 mg on day 1 and at weeks 4 and 8 by subcutaneous injection during the double-blind treatment phase.
  In the open-label treatment phase participants received 70 mg erenumab QM from week 12 to week 264 (last dose). After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
  Interventions: Drug: Erenumab
- Erenumab 70 mg QM (Experimental): Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection during the double-blind treatment phase.
  In the open-label treatment phase participants received 70 mg erenumab QM from week 12 to week 264 (last dose). After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
  Interventions: Drug: Erenumab
- CHU Substudy: Erenumab 140 mg PFS (Experimental): Participants in the open-label treatment phase in the United States randomized to self-administer 140 mg erenumab via two 70 mg injections using a prefilled syringe (PFS) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
  Interventions: Drug: Erenumab PFS
- CHU Substudy: Erenumab 140 mg AI/Pen (Experimental): Participants in the open-label treatment phase in the United States randomized to self-administer 140 mg erenumab via two 70 mg injections using an autoinjector/pen (AI)/pen) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
  Interventions: Drug: Erenumab AI/Pen

INTERVENTIONS:
Drug: Erenumab — Administered by study site staff once a month (QM) as a subcutaneous injection
  Other Names: AMG 334; Aimovig™
  Arms: Erenumab 21 mg QM; Erenumab 7 mg QM; Erenumab 70 mg QM; Placebo
Drug: Placebo — Administered by study site staff once a month (QM) as a subcutaneous injection
  Arms: Placebo
Drug: Erenumab PFS — Erenumab supplied in a single-use prefilled syringe for self-administration in the CHU substudy
  Arms: CHU Substudy: Erenumab 140 mg PFS
Drug: Erenumab AI/Pen — Erenumab supplied in a single-use autoinjector/pen for self-administration in the CHU substudy
  Arms: CHU Substudy: Erenumab 140 mg AI/Pen

SUMMARY:
A study to evaluate the effect of erenumab compared to placebo on the change from baseline in monthly migraine days in participants with episodic migraine.

DETAILED DESCRIPTION:
The study is composed of an initial screening phase (up to 3 weeks), a 4-week baseline phase, a 12-week double-blind treatment phase (DBTP), an open-label treatment phase (OLTP) for up to 256 weeks, and an 8-week safety follow-up (12 weeks after the last dose of investigational product [IP]).

In the DBTP participants were to be randomized in a 3:2:2:2 ratio to placebo, erenumab 7 mg, erenumab 21 mg, or erenumab 70 mg.

During the open-label treatment phase, participants were to receive erenumab 70 mg QM from week 12 to week 264. After implementation of Protocol Amendment 3 (07 April 2016), participants remaining in the OLTP increased their dose to erenumab 140 mg QM up to week 264. The safety follow-up increased from an 8-week safety follow-up to a 12-week safety follow-up (16 weeks after the last dose of investigational product).

During the OLTP participants enrolled at sites in the United States could enroll in an optional clinical home use (CHU) substudy, per a country-specific protocol amendment dated 20 June 2016. Participants in the CHU substudy were to be randomized 1:1 into 1 of 2 treatment groups: erenumab 140 mg using a prefilled syringe or erenumab 140 mg using an autoinjector/pen. Day 1 of the CHU substudy corresponded with any OLTP study visit up through Week 256, as long as the participant had received at least 2 doses of erenumab 140 mg. During the CHU substudy, participants initially self-administered IP under site supervision on substudy day 1, and then self-administered IP at home on substudy days 29 and 57.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine for more than12 months prior to screening
* Migraine frequency: ≥ 4 and ≤ 14 migraine days per month in each of the 3 months prior to screening and during baseline phase
* Headache frequency: < 15 headache days per month (with > 50% of the headache days being migraine days) in each of the 3 months prior to screening and during baseline phase
* Demonstrated at least 80% compliance with the eDiary during baseline phase

Exclusion Criteria:

* Older than 50 years of age at migraine onset
* History of cluster headache or basilar or hemiplegic migraine headache
* Unable to differentiate migraine from other headaches
* No therapeutic response with > 2 of the following eight medication categories for prophylactic treatment of migraine after an adequate therapeutic trial. Medication categories are:

  * Category 1: Divalproex sodium, sodium valproate
  * Category 2: Topiramate
  * Category 3: Beta blockers (for example: atenolol, bisoprolol, metoprolol, nadolol, nebivolol, pindolol, propranolol, timolol)
  * Category 4: Tricyclic antidepressants (for example: amitriptyline, nortriptyline, protriptyline)
  * Category 5: Venlafaxine, desvenlafaxine, duloxetine, milnacipran
  * Category 6: Flunarizine, verapamil
  * Category 7: Lisinopril, candesartan
  * Category 8: Butterbur, feverfew, magnesium (≥ 600 mg/day), riboflavin (≥ 100 mg/day)
* Overuse of acute migraine medications in any month during the 3 months prior to screening or during screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 483 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2014-09-25 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (61):
- United States (39):
  - Research Site, Phoenix, Arizona
  - Research Site, Long Beach, California
  - Research Site, National City, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Spring Valley, California
  - Research Site, Danbury, Connecticut
  - Research Site, Fairfield, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Watertown, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Plymouth, Minnesota
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Rochester, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Falls Church, Virginia
  - Research Site, Virginia Beach, Virginia
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Denmark (2):
  - Research Site, Aarhus C
  - Research Site, Glostrup Municipality
- Finland (5):
  - Research Site, Helsinki
  - Research Site, Mikkeli
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- Germany (5):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Leipzig
- Norway (4):
  - Research Site, Ålesund
  - Research Site, Hamar
  - Research Site, Sandvika
  - Research Site, Stavanger
- Sweden (4):
  - Research Site, Falköping
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Vällingby

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Sun H, Dodick DW, Silberstein S, Goadsby PJ, Reuter U, Ashina M, Saper J, Cady R, Chon Y, Dietrich J, Lenz R. Safety and efficacy of AMG 334 for prevention of episodic migraine: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Apr;15(4):382-90. doi: 10.1016/S1474-4422(16)00019-3. Epub 2016 Feb 12. PMID 26879279
- [Background] Ashina M, Dodick D, Goadsby PJ, Reuter U, Silberstein S, Zhang F, Gage JR, Cheng S, Mikol DD, Lenz RA. Erenumab (AMG 334) in episodic migraine: Interim analysis of an ongoing open-label study. Neurology. 2017 Sep 19;89(12):1237-1243. doi: 10.1212/WNL.0000000000004391. Epub 2017 Aug 23. PMID 28835404
- [Background] Ashina M, Goadsby PJ, Reuter U, Silberstein S, Dodick D, Rippon GA, Klatt J, Xue F, Chia V, Zhang F, Cheng S, Mikol DD. Long-term safety and tolerability of erenumab: Three-plus year results from a five-year open-label extension study in episodic migraine. Cephalalgia. 2019 Oct;39(11):1455-1464. doi: 10.1177/0333102419854082. Epub 2019 May 30. PMID 31146544
- [Background] Cheng S, Picard H, Zhang F, Eisele O, Mikol DD. Efficacy and safety of erenumab for migraine prevention: an overview. Japanese Journal of Headache. 2019; 45 : 493-505.
- [Background] Ashina M, Goadsby PJ, Reuter U, Silberstein S, Dodick DW, Xue F, Zhang F, Paiva da Silva Lima G, Cheng S, Mikol DD. Long-term efficacy and safety of erenumab in migraine prevention: Results from a 5-year, open-label treatment phase of a randomized clinical trial. Eur J Neurol. 2021 May;28(5):1716-1725. doi: 10.1111/ene.14715. Epub 2021 Jan 20. PMID 33400330
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Ashina M, Kudrow D, Reuter U, Dolezil D, Silberstein S, Tepper SJ, Xue F, Picard H, Zhang F, Wang A, Zhou Y, Hong F, Klatt J, Mikol DD. Long-term tolerability and nonvascular safety of erenumab, a novel calcitonin gene-related peptide receptor antagonist for prevention of migraine: A pooled analysis of four placebo-controlled trials with long-term extensions. Cephalalgia. 2019 Dec;39(14):1798-1808. doi: 10.1177/0333102419888222. Epub 2019 Nov 10. PMID 31707815
- [Background] Kudrow D, Pascual J, Winner PK, Dodick DW, Tepper SJ, Reuter U, Hong F, Klatt J, Zhang F, Cheng S, Picard H, Eisele O, Wang J, Latham JN, Mikol DD. Vascular safety of erenumab for migraine prevention. Neurology. 2020 Feb 4;94(5):e497-e510. doi: 10.1212/WNL.0000000000008743. Epub 2019 Dec 18. PMID 31852816
- [Background] Sakai F, Takeshima T, Tatsuoka Y, Hirata K, Cheng S, Numachi Y, Peng C, Xue F, Mikol DD. Long-term efficacy and safety during open-label erenumab treatment in Japanese patients with episodic migraine. Headache. 2021 Apr;61(4):653-661. doi: 10.1111/head.14096. Epub 2021 Mar 25. PMID 33764538
- [Derived] Ashina M, Goadsby PJ, Dodick DW, Tepper SJ, Xue F, Zhang F, Brennan F, Paiva da Silva Lima G. Assessment of Erenumab Safety and Efficacy in Patients With Migraine With and Without Aura: A Secondary Analysis of Randomized Clinical Trials. JAMA Neurol. 2022 Feb 1;79(2):159-168. doi: 10.1001/jamaneurol.2021.4678. PMID 34928306
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 59 centers in North America (Canada, USA) and Europe (Denmark, Finland, Germany, Norway, Sweden, and Portugal).
  The study consisted of a 12-week double-blind treatment phase (DBTP) and a 256-week open-label treatment phase (OLTP) followed by a safety follow-up of 8 to 12 weeks (12 -16 weeks after last dose). The OLTP portion of the study was not conducted in Norway.
Pre-assignment Details: Participants were randomized 3:2:2:2 to receive placebo, erenumab 7 mg, erenumab 21 mg, or erenumab 70 mg once a month (QM) in the double-blind phase. Randomization was stratified by region (North America vs. Europe).
  During the open-label treatment phase, participants in the United States (US) could participate in an optional Clinical Home Use (CHU) substudy.
Groups:
- DBTP: Placebo QM: Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- DBTP: Erenumab 7 mg QM: Participants received erenumab 7 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- DBTP: Erenumab 21 mg QM: Participants received erenumab 21 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- DBTP: Erenumab 70 mg QM: Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- OLTP: Erenumab 70/140 mg QM: Participants received 70 mg erenumab QM from the beginning of the OLTP (week 12). After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
- CHU Substudy: Erenumab 140 mg by Prefilled Syringe: Participants in the open-label treatment phase in the United States randomized to self-administer 140 mg erenumab via two 70 mg injections using a prefilled syringe (PFS) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
- CHU Substudy: Erenumab 140 mg Autoinjector/Pen: Participants in the open-label treatment phase in the United States randomized to self-administer 140 mg erenumab via two 70 mg injections using an autoinjector (AI)/pen on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
Period: Double-blind Treatment Phase
Arm/Group | DBTP: Placebo QM | DBTP: Erenumab 7 mg QM | DBTP: Erenumab 21 mg QM | DBTP: Erenumab 70 mg QM | OLTP: Erenumab 70/140 mg QM | CHU Substudy: Erenumab 140 mg by Prefilled Syringe | CHU Substudy: Erenumab 140 mg Autoinjector/Pen
Started | 160 | 108 | 108 | 107 | 0 | 0 | 0
Received Study Drug | 153 | 108 | 105 | 106 | 0 | 0 | 0
Completed (Completed double-blind treatment phase) | 143 | 105 | 99 | 101 | 0 | 0 | 0
Not Completed | 17 | 3 | 9 | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 3 | 3 | 4 | 0 | 0 | 0
Not completed — Sponsor Decision | 6 | 0 | 5 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 0 | 0
Period: Open-label Treatment Phase
Arm/Group | DBTP: Placebo QM | DBTP: Erenumab 7 mg QM | DBTP: Erenumab 21 mg QM | DBTP: Erenumab 70 mg QM | OLTP: Erenumab 70/140 mg QM | CHU Substudy: Erenumab 140 mg by Prefilled Syringe | CHU Substudy: Erenumab 140 mg Autoinjector/Pen
Started (Participants enrolled in Norway did not participate in the OLTP. In addition 12 participants who completed the DBTP withdrew consent prior to entering the OLTP.) | 0 | 0 | 0 | 0 | 383 | 0 | 0
Received 70 mg Erenumab | 0 | 0 | 0 | 0 | 383 | 0 | 0
Received 140 mg Erenumab | 0 | 0 | 0 | 0 | 250 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 221 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 162 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 121 | 0 | 0
Not completed — Decision by Sponsor | 0 | 0 | 0 | 0 | 17 | 0 | 0
Not completed — Missing | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 19 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Clinical Home Use Substudy
Arm/Group | DBTP: Placebo QM | DBTP: Erenumab 7 mg QM | DBTP: Erenumab 21 mg QM | DBTP: Erenumab 70 mg QM | OLTP: Erenumab 70/140 mg QM | CHU Substudy: Erenumab 140 mg by Prefilled Syringe | CHU Substudy: Erenumab 140 mg Autoinjector/Pen
Started | 0 | 0 | 0 | 0 | 0 | 42 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 39 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Decision by Sponsor | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- Erenumab 7 mg QM: Participants received erenumab 7 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- Erenumab 21 mg QM: Participants received erenumab 21 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- Erenumab 70 mg QM: Participants received erenumab 70 mg on day 1 and at weeks 4 and 8 by subcutaneous injection in the double-blind treatment phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Erenumab 7 mg QM | Erenumab 21 mg QM | Erenumab 70 mg QM | Total
Number analyzed (Participants) | 160 | 108 | 108 | 107 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (10.0) | 40.3 (10.9) | 39.9 (12.3) | 42.6 (9.9) | 41.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 88 | 87 | 82 | 389
  Male | 28 | 20 | 21 | 25 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 9 | 1 | 30
  Not Hispanic or Latino | 149 | 99 | 99 | 106 | 453
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 1 | 4
  Black or African American | 13 | 10 | 7 | 2 | 32
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White | 142 | 97 | 100 | 103 | 442
  Multiple | 0 | 0 | 0 | 1 | 1
  Other | 2 | 1 | 0 | 0 | 3
Region [Count of Participants; unit: Participants] — Region is based on actual data collected at study baseline instead of randomization stratification.
  Participants
    North America | 85 | 58 | 58 | 58 | 259
    Europe | 75 | 50 | 50 | 49 | 224
Monthly Migraine Days [Mean (Standard Deviation); unit: migraine days/month] — A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase. Population: Participants with available baseline data
  migraine days/month
    number analyzed (Participants) | 160 | 108 | 108 | 106 | 482
    (all) | 8.77 (2.72) | 8.62 (2.79) | 8.93 (2.88) | 8.58 (2.49) | 8.73 (2.72)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days at Week 12
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura. The change from baseline in monthly migraine days was calculated as the number of migraine days during the last 4 weeks of the 12-week double-blind treatment phase - the number of migraine days during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: Participants who received at least 1 dose of investigational product (IP) and had ≥ 4 migraine days during the 4-week baseline phase (efficacy analysis set), and with at least one change from baseline value in monthly migraine days.
Measure: Least Squares Mean (Standard Error); unit: migraine days / month
Arm/Group | Placebo | Erenumab 7 mg QM | Erenumab 21 mg QM | Erenumab 70 mg QM
Number analyzed (Participants) | 152 | 107 | 99 | 104
migraine days / month | -2.28 (0.31) | -2.18 (0.36) | -2.39 (0.38) | -3.40 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; The primary analysis utilized a generalized linear mixed model which included treatment, visit, treatment by visit, the stratification factor region, and baseline value as covariates; Test type: Superiority — To maintain the type I error at ≤ 0.05, the pairwise comparison was tested in a sequential testing procedure in the order of erenumab 70 mg vs placebo, 21 mg vs placebo, and 7 mg vs placebo. The lower dose group was only to be tested when the higher dose group was tested as significant; p = 0.021, Generalized Linear Mixed Model; LS Mean Difference = -1.12, 95% CI 2-sided [-2.06 to -0.17]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 21 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.83, Generalized Linear Mixed Model; LS Mean Difference = -0.10, 95% CI 2-sided [-1.07 to 0.86]
Statistical Analysis 3: Comparison: Placebo vs Erenumab 7 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.82, Generalized Linear Mixed Model; LS Mean Difference = 0.11, 92% CI 2-sided [-0.83 to 1.05]

2. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Monthly Migraine Days at Week 12
Description: A migraine day was any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache was defined either as a migraine without aura or a migraine with aura. Monthly migraine days were calculated as the number of migraine days in the 4-week baseline phase and during the last 4 weeks of double-blind treatment. At least a 50% reduction from baseline in monthly migraine days was determined if the change in monthly migraine days from the 4-week baseline phase to the last 4 weeks of the 12-week double-blind treatment phase * 100 / baseline monthly migraine days was less than or equal to -50%.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: Participants who received at least 1 dose of investigational product and had ≥ 4 migraine days during the 4-week baseline phase (efficacy analysis set) with available data at week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Erenumab 7 mg QM | Erenumab 21 mg QM | Erenumab 70 mg QM
Number analyzed (Participants) | 144 | 104 | 93 | 99
percentage of participants | 29.9 | 28.8 | 34.4 | 46.5
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; The generalized linear mixed model includes data for all participants in the efficacy analysis set with at least one percent change from baseline value in monthly migraine days (152 participants in the placebo group and 104 in the erenumab 70 mg group); Test type: Superiority; p = 0.011, Generalised Linear Mixed Model; Generalized linear mixed model including treatment, visit, treatment by visit, stratification factor region, and baseline value as covariates; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.17 to 3.42]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 21 mg QM; The generalized linear mixed model includes data for all participants in the efficacy analysis set with at least one change from baseline value in monthly migraine days (152 participants in the placebo group and 99 in the erenumab 21 mg group); Test type: Superiority; p = 0.44, Generalized Linear Mixed Model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.71 to 2.18]
Statistical Analysis 3: Comparison: Placebo vs Erenumab 7 mg QM; The generalized linear mixed model includes data for all participants in the efficacy analysis set with at least one change from baseline value in monthly migraine days (152 participants in the placebo group and 107 in the erenumab 7 mg group); Test type: Superiority; p = 0.80, Generalized Linear Mixed Model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.53 to 1.63]

3. Secondary Outcome: Change From Baseline in Monthly Migraine Attacks at Week 12
Description: A migraine attack is an episode of any qualified migraine headache or migraine specific medication intakes for aura only. A migraine attack that was interrupted by sleep or that temporarily remits and then recurs within 48 hours or an attack treated successfully with medication but that relapses within 48 hours was considered to be one attack.
  The change from baseline in monthly migraine attacks was calculated as the number of migraine attacks during the last 4 weeks of the 12-week double-blind treatment phase - the number of migraine attacks during the 4-week baseline phase.
Time Frame: 4-week baseline phase and the last 4 weeks of the 12-week double-blind treatment phase
Population: Participants who received at least 1 dose of investigational product and had ≥ 4 migraine days during the 4-week baseline phase (efficacy analysis set), and with at least one change from baseline value in monthly migraine attacks.
Measure: Least Squares Mean (Standard Error); unit: migraine attacks/month
Arm/Group | Placebo | Erenumab 7 mg QM | Erenumab 21 mg QM | Erenumab 70 mg QM
Number analyzed (Participants) | 152 | 107 | 99 | 104
migraine attacks/month | -1.44 (0.17) | -1.07 (0.20) | -1.42 (0.21) | -1.84 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Erenumab 70 mg QM; Test type: Superiority; p = 0.13, Generalized Linear Mixed Model; Generalized linear mixed model including treatment, visit, treatment by visit, the stratification factor region, and baseline value as covariates; LS Mean Difference = -0.40, 95% CI 2-sided [-0.92 to 0.12]
Statistical Analysis 2: Comparison: Placebo vs Erenumab 21 mg QM; Test type: Superiority; p = 0.95, Generalized Linear Mixed Model; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = 0.02, 95% CI 2-sided [-0.51 to 0.54]
Statistical Analysis 3: Comparison: Placebo vs Erenumab 7 mg QM; Test type: Superiority; p = 0.16, Generalized Linear Mixed Model; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = 0.37, 95% CI 2-sided [-0.14 to 0.87]

4. Primary Outcome: CHU Substudy: Number of Participants Who Self-administered a Full Dose, Partial Dose, or No Dose of Erenumab
Description: To assess participants ability to administer a full dose of erenumab in home-use at day 29 (week 4) and day 57 (week 8), site staff called participants and asked whether the participant administered a full, partial, or no dose of erenumab. A full dose means that the entire volume of both prefilled syringes or autoinjector/pens were injected. Discontinued prior to dosing day indicates participants who had discontinued the investigational product and did not attempt to self-administer on day 29 or 57.
Time Frame: CHU substudy day 29 (week 4) and day 57 (week 8)
Population: Participants enrolled in the CHU substudy who received at least 1 dose of investigational product in the substudy.
Measure: Count of Participants; unit: Participants
Groups:
- CHU Substudy: Erenumab 140 mg Prefilled Syringe: Participants in the open-label treatment phase in the United States self-administered 140 mg erenumab via two 70 mg injections using a prefilled syringe (PFS) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
- CHY SubStudy: Erenumab 140 mg Autoinjector/Pen: Participants in the open-label treatment phase in the United States self-administered 140 mg erenumab via two 70 mg injections using an autoinjector/pen (AI)/pen) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
Arm/Group | CHU Substudy: Erenumab 140 mg Prefilled Syringe | CHY SubStudy: Erenumab 140 mg Autoinjector/Pen
Number analyzed (Participants) | 42 | 41
Participants
  Day 29 (week 4): Full dose | 39 | 41
  Day 29 (week 4): Partial dose | 1 | 0
  Day 29 (week 4): Discontinued prior to dosing day | 2 | 0
  Day 57 (week 8): Full dose | 39 | 39
  Day 57 (week 8): Partial dose | 0 | 1
  Day 57 (week 8): Discontinued prior to dosing day | 3 | 1

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events in the Double-blind Treatment Phase
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial subject, including worsening of a pre-existing medical condition and laboratory value changes that require treatment or adjustment in current therapy.
  AEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03:
  1. Mild; asymptomatic or mild symptoms
  2. Moderate; minimal, local or noninvasive intervention indicated; limiting daily activities
  3. Severe or medically significant but not immediately life-threatening; hospitalization indicated; disabling; limiting self-care
  4. Life-threatening consequences; urgent intervention indicated
  5. Death related to AE
  A serious adverse event is an AE that meets at least 1 of the following criteria:
  * fatal
  * life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
Time Frame: From first dose of study drug in the double-blind treatment phase until the first dose of study drug in the open-label treatment phase (12 weeks) or up to 12 weeks after last dose for participants who did not enter the open-label treatment phase.
Population: Randomized participants who received at least one dose of investigational product (safety analysis set).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab 7 mg QM | Erenumab 21 mg QM | Erenumab 70 mg QM
Number analyzed (Participants) | 153 | 108 | 105 | 106
Participants
  Any adverse event (AE) | 81 | 57 | 55 | 57
  Serious adverse events (SAEs) | 1 | 1 | 0 | 1
  AE leading to discontinuation of IP | 2 | 2 | 2 | 3
  AE Grade ≥ 2 | 36 | 31 | 25 | 23
  AE Grade ≥ 3 | 3 | 3 | 3 | 3
  AE Grade ≥ 4 | 0 | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events in the Open-label Treatment Phase
Description: as for outcome 5
Time Frame: From first dose in the open-label treatment phase up to 12 weeks (participants receiving 70 mg only) or 16 weeks (participants with dose increased to 140 mg) after the last dose; a maximum of 268 weeks.
Population: All participants who received at least one dose of investigational product in the open-label treatment phase (open-label treatment phase set).
Measure: Count of Participants; unit: Participants
Groups:
- OLTP: Erenumab 70 mg QM: Participants received 70 mg erenumab QM from week 12 until implementation of Protocol Amendment 3 (07 April 2016) in the open-label treatment phase; median duration of exposure was 104 weeks.
- OLTP: Erenumab 140 mg QM: After implementation of Protocol Amendment 3 (07 April 2016), participants still on study received erenumab 140 mg QM up to week 264 in the open-label treatment phase; median duration of exposure was 141 weeks.
Arm/Group | OLTP: Erenumab 70 mg QM | OLTP: Erenumab 140 mg QM | OLTP: Erenumab 70/140 mg QM
Number analyzed (Participants) | 383 | 250 | 383
Participants
  Any adverse event (AE) | 323 | 216 | 340
  Serious adverse events (SAEs) | 30 | 25 | 49
  AE leading to discontinuation of IP | 16 | 2 | 18
  AE Grade ≥ 2 | 249 | 180 | 286
  AE Grade ≥ 3 | 55 | 40 | 83
  AE Grade ≥ 4 | 1 | 3 | 4
  Fatal adverse events | 1 | 1 | 2

7. Secondary Outcome: CHU Substudy: Number of Participants With Treatment-emergent Adverse Events During the CHU Substudy
Description: AEs were graded using the CTCAE version 4.03:
  1. Mild; asymptomatic or mild symptoms
  2. Moderate; minimal, local or noninvasive intervention indicated; limiting daily activities
  3. Severe or medically significant but not immediately life-threatening; hospitalization indicated; disabling; limiting self-care
  4. Life-threatening consequences; urgent intervention indicated
  5. Death related to AE
  A serious adverse event is an AE that meets at least 1 of the following criteria:
  * fatal
  * life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event An adverse device effect is any AE related to the use of a medical device, including AEs resulting from insufficient or inadequate instructions for use, any malfunction of the device, or use error or from intentional misuse of the device.
Time Frame: From first dose in the CHU substudy to end of substudy (up to 12 weeks)
Population: Participants enrolled in the CHU substudy who received at least 1 dose of investigational product in the substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | CHU Substudy: Erenumab 140 mg Prefilled Syringe | CHY SubStudy: Erenumab 140 mg Autoinjector/Pen
Number analyzed (Participants) | 42 | 41
Participants
  Any adverse event | 13 | 17
  AE Grade ≥ 2 | 7 | 10
  AE Grade ≥ 3 | 1 | 2
  AE Grade ≥ 4 | 0 | 0
  Serious adverse events | 0 | 0
  Leading to discontinuation of IP | 0 | 0
  Fatal adverse events | 0 | 0
  Injection site reactions | 4 | 2
  Adverse device effects | 2 | 2

8. Secondary Outcome: Number of Participants Who Developed Anti-erenumab Antibodies During the Double-blind Treatment Phase
Description: Two validated assays were used to detect the presence of anti-erenumab antibodies. First, an electrochemiluminescent bridging immunoassay was used to detect binding antibodies (screening assay) and confirm antibodies (confirmatory assay) capable of binding erenumab. Second, a cell-based bioassay was used to test positive binding antibody samples for neutralizing activity against erenumab.
  Participants who developed anti-erenumab antibodies are participants who were negative or had no result at baseline but positive at any time postbaseline during the DBTP.
  If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the participant was defined as positive for neutralizing antibodies.
Time Frame: 12 weeks
Population: Participants who received at least 1 dose of IP and with valid postbaseline antibody testing results.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Erenumab 7 mg QM | Erenumab 21 mg QM | Erenumab 70 mg QM
Number analyzed (Participants) | 149 | 107 | 104 | 106
Participants
  Developed binding antibodies | 0 | 13 | 12 | 8
  Developed neutralizing antibodies | 0 | 5 | 3 | 1

9. Secondary Outcome: Number of Participants Who Developed Anti-erenumab Antibodies During the Open-label Treatment Phase
Description: Two validated assays were used to detect the presence of anti-erenumab antibodies. First, an electrochemiluminescent bridging immunoassay was used to detect binding antibodies (screening assay) and confirm antibodies (confirmatory assay) capable of binding erenumab. Second, a cell-based bioassay was used to test positive binding antibody samples for neutralizing activity against erenumab.
  Participants who developed anti-erenumab antibodies are participants who were negative prior to the first OLTP dose but positive at any time during the OLTP, or participants with no data prior to first dose in OLTP with any post-baseline positive results.
  If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the participant was defined as positive for neutralizing antibodies.
Time Frame: From week 12 up to 12 weeks (participants receiving 70 mg only) or 16 weeks (participants with dose increased to 140 mg) after the last dose; maximum 268 weeks.
Population: Participants who received at least 1 dose of IP in the OLTP and with valid antibody testing results during the OLTP.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo / Erenumab 70/140 mg QM: Participants randomized to placebo in the double-blind treatment phase received 70 mg erenumab QM from week 12 in the open-label treatment phase. After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
- Erenumab 7 mg QM / Erenumab 70/140 mg QM: Participants randomized to erenumab 7 mg in the double-blind treatment phase received 70 mg erenumab QM from week 12 in the open-label treatment phase. After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
- Erenumab 21 mg QM / Erenumab 70/140 mg QM: Participants randomized to erenumab 21 mg in the double-blind treatment phase received 70 mg erenumab QM from week 12 in the open-label treatment phase. After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
- Erenumab 70 mg QM / Erenumab 70/140 mg QM: Participants randomized to erenumab 70 mg in the double-blind treatment phase received 70 mg erenumab QM from week 12 in the open-label treatment phase. After Protocol Amendment 3, participants still on study had their dose increased to 140 mg QM.
Arm/Group | Placebo / Erenumab 70/140 mg QM | Erenumab 7 mg QM / Erenumab 70/140 mg QM | Erenumab 21 mg QM / Erenumab 70/140 mg QM | Erenumab 70 mg QM / Erenumab 70/140 mg QM
Number analyzed (Participants) | 119 | 88 | 87 | 86
Participants
  Developed binding antibodies | 12 | 8 | 6 | 5
  Developed neutralizing antibodies | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Double-blind Treatment Phase: From first dose of study drug in the DBTP until the first dose of study drug in the open-label treatment phase (12 weeks) or up to 12 weeks after last dose for participants who did not enter the open-label treatment phase. Open-label Treatment Phase: From first dose in the OLTP up to 12 weeks (participants receiving 70 mg only) or 16 weeks (participants with dose increased to 140 mg) after the last dose; maximum 268 weeks. CHU substudy: 12 weeks
Groups:
- CHU Substudy: Erenumab 140 mg PFS: Participants in the open-label treatment phase in the United States self-administered 140 mg erenumab via two 70 mg injections using a prefilled syringe (PFS) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
- CHU Substudy: Erenumab 140 mg AI/Pen: Participants in the open-label treatment phase in the United States self-administered 140 mg erenumab via two 70 mg injections using an autoinjector/pen (AI)/pen) on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
- CHU Substudy: Total: Participants in the open-label treatment phase in the United States self-administered 140 mg erenumab via two 70 mg injections using a prefilled syringe or autoinjector/pen on CHU substudy day 1 (under study site supervision), and at home on day 29 (week 4) and day 57 (week 8).
Arm/Group | DBTP: Placebo QM | DBTP: Erenumab 7 mg QM | DBTP: Erenumab 21 mg QM | DBTP: Erenumab 70 mg QM | OLTP: Erenumab 70 mg QM | OLTP: Erenumab 140 mg QM | OLTP: Erenumab 70/140 mg QM | CHU Substudy: Erenumab 140 mg PFS | CHU Substudy: Erenumab 140 mg AI/Pen | CHU Substudy: Total
Serious Adverse Events (participants affected / at risk) | 1/153 | 1/108 | 0/105 | 1/106 | 30/383 | 25/250 | 49/383 | 0/42 | 0/41 | 0/83
Other Adverse Events (participants affected / at risk) | 45/153 | 27/108 | 24/105 | 31/106 | 220/383 | 172/250 | 264/383 | 7/42 | 9/41 | 16/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBTP: Placebo QM (N=153) | DBTP: Erenumab 7 mg QM (N=108) | DBTP: Erenumab 21 mg QM (N=105) | DBTP: Erenumab 70 mg QM (N=106) | OLTP: Erenumab 70 mg QM (N=383) | OLTP: Erenumab 140 mg QM (N=250) | OLTP: Erenumab 70/140 mg QM (N=383) | CHU Substudy: Erenumab 140 mg PFS (N=42) | CHU Substudy: Erenumab 140 mg AI/Pen (N=41) | CHU Substudy: Total (N=83)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Primary hyperaldosteronism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Appendicitis noninfective (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBTP: Placebo QM (N=153) | DBTP: Erenumab 7 mg QM (N=108) | DBTP: Erenumab 21 mg QM (N=105) | DBTP: Erenumab 70 mg QM (N=106) | OLTP: Erenumab 70 mg QM (N=383) | OLTP: Erenumab 140 mg QM (N=250) | OLTP: Erenumab 70/140 mg QM (N=383) | CHU Substudy: Erenumab 140 mg PFS (N=42) | CHU Substudy: Erenumab 140 mg AI/Pen (N=41) | CHU Substudy: Total (N=83)
Nasopharyngitis (Infections and infestations) | 12 | 10 | 6 | 6 | 82 | 59 | 111 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 9 | 15 | 24 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 13 | 18 | 29 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 5 | 2 | 4 | 19 | 11 | 29 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 17 | 14 | 31 | 0 | 0 | 0
Influenza (Infections and infestations) | 5 | 1 | 4 | 1 | 36 | 31 | 56 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 11 | 11 | 22 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 1 | 2 | 30 | 26 | 53 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2 | 2 | 52 | 53 | 78 | 3 | 2 | 5
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 23 | 23 | 41 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 1 | 26 | 13 | 37 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4 | 2 | 30 | 21 | 48 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 16 | 11 | 25 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 1 | 3 | 10 | 11 | 21 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 15 | 14 | 27 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 15 | 7 | 20 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 0 | 2 | 14 | 11 | 25 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.